CLINICAL TRIAL: NCT00038935
Title: A Single Dose, Randomized, Double-Blind, 2-Period Crossover Study in Patients With Hemophilia A to Evaluate the Pharmacokinetics of B-Domain Deleted Recombinant Human Factor VIII (BDDrFVIII) Manufactured by the Current Process (ReFacto) and by an Albumin Free Manufacturing Process (ReFacto AF)
Brief Title: Study Evaluating BDDRFVIII and ReFacto AF in Hemophilia A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3082B1-305
Record Dates: First submitted 2002-06-05; First posted 2002-06-07 (Estimated); Last update posted 2008-04-22 (Estimated); Status verified 2008-04

CONDITIONS: Hemophilia A
Keywords: Hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

INTERVENTIONS:
Drug: ReFacto AF

SUMMARY:
The purpose of this study is to determine the relative bioavailability of ReFacto AF as compared to ReFacto, when each is administered as 2-minute bolus infusions.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A (FVIII:C < 1% at local laboratory)
* Previously treated patients (PTP) with at least 250 exposure days to any factor VIII product
* Age greater than or equal to 12 years\

Exclusion Criteria:

* The presence of any bleeding disorder in addition to hemophilia A
* Concomitant therapy with immunosuppressant drugs (e.g., intravenous immunoglobulin (IVIG), routine systemic corticosteroid use)
* History of detectable factor VIII inhibitor

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Korth-Bradley J, Rupon J, Plotka A, Charnigo R, Rendo P. Assessment of Relative Bioavailability of Moroctocog Alfa and Moroctocog Alfa (AF-CC) in Subjects With Severe Hemophilia A. Clin Transl Sci. 2018 May;11(3):283-288. doi: 10.1111/cts.12544. Epub 2018 Mar 25. PMID 29575770